CLINICAL TRIAL: NCT05371639
Title: Efficacy and Safety of Tian Ma Bian Chun Zhi Gan Tablets in the Treatment of Mild to Moderate Vascular Dementia: a Randomized, Placebo Controlled, Double Blind, Parallel Group, Multicenter Trial
Brief Title: Efficacy and Safety of Tian Ma Bian Chun Zhi Gan Tablets in Mild to Moderate Vascular Dementia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Doctor, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YHNK-XY-2-2021-01
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Vascular Dementia; Cognitive Impairment
Keywords: Vascular dementia; Cognitive impairment; Tian Ma Bian Chun Zhi Gan; Randomized clinical trial
MeSH Terms: conditions — Dementia, Vascular; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tian Ma Bian Chun Zhi Gan group (Experimental): Tian Ma Bian Chun Zhi Gan tablets
  Interventions: Drug: Tian Ma Bian Chun Zhi Gan Tablets
- Placebo group (Placebo Comparator): placebo identified to Tian Ma Bian Chun Zhi Gan tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tian Ma Bian Chun Zhi Gan Tablets — Tian Ma Bian Chun Zhi Gan Tablets, 0.1g per pill which contains 14mg Tian Ma Bian Chun Zhi Gan, 3 pills per time, 2 times per day for 36 weeks.
  Arms: Tian Ma Bian Chun Zhi Gan group
Drug: Placebo — Placebo identified to Tian Ma Bian Chun Zhi Gan, 0.1g per pill which contains 0mg Tian Ma Bian Chun Zhi Gan, 3 pills per time, 2 times per day for 36 weeks.
  Arms: Placebo group

SUMMARY:
The study will be a 36-week multicentre, double-blind, placebo-controlled phase Ⅱb trial in China. Total 360 participants aged 55-80 years will be randomized to Tian Ma Bian Chun Zhi Gan group (84mg per day) or to placebo group. The primary endpoint will be Vascular Dementia Assessment Scale-cognitive subscale and Clinical Dementia Rating-Sum of Boxes. Secondary outcomes included changes in Mini-Mental State Examination, Clock Drawing Test, Delayed Story Recall and Ability of Daily Living. Patients' safety will be assessed by recording of adverse events, clinical examinations, electrocardiography and laboratory tests. The patients, caregivers, and investigators will be blinded to the treatment allocations.

ELIGIBILITY:
Inclusion Criteria:

1. Concerns of a patient, knowledgeable informant or a clinician of decline from a previous level of cognitive functioning.
2. Clear and significant deficits in objective assessment in two or more cognitive domains, Memory decline, delayed story recall ≤10.5point(maximum is 56 point), or visuoconstructional-perceptual ability, clock drawing test≤3point(maximum is 4 point);or executive function, trail making test-part B≥188.5 second( maximun is 300 second); or language function, boston naming test-30 items ≤21.5 point( maximum is 30);
3. Global cognitive impairment, mild to moderate dementia with Mini-mental state examination(MMSE) score of ≤26 and ≥11;
4. Cognitive deficits are severe enough to impair social or occupational functioning, the ability of daily living scale ≥16 points;
5. Determining evidence of significant cerebrovascular disease, presence of significant neuroimaging (MRI or CT) evidence of cerebrovascular disease (one of the following): a) multiple (≥2) large vessel infarcts ; b) Single lacunes placed strategically in the thalamus or basal ganglia; c) Multiple lacunar infarcts (≥3) outside the brainstem; d) 1-2 lacunes may be sufficient if strategically placed or in combination with extensive white matter lesions; e) extensive and confluent white matter lesions; f) watershed infarction with moderate white matter lesions; g) Strategically placed intracerebral hemorrhage, or two or more intracerebral hemorrhages; h) combination of the above.
6. A relationship between dementia and cerebro-vascular disease, manifested or inferred by the presence of one or more of the following: a) abrupt deterioration in cognitive functions, the onset of the cognitive deficits is temporally related to one or more cerebro-vascular events , onset of cognitive deficits within 3 months following a recognized stroke, and cognitive deficits persisting beyond three months after the event, and abrupt with a stepwise or fluctuating course owing to multiple such events; b) gradual onset and slowly progressive course, evidence for decline is prominent in speed of information processing, complex attention and/or frontal-executive functioning in the absence of history of a stroke or transient ischemic attack. One of the following features is additionally present: ①Early presence of a gait disturbance; ②Early urinary frequency, urgency, and other urinary symptoms not explained by urologic disease; ③Personality and mood changes: abulia, depression, or emotional incontinence
7. Aged ≥55 and ≤80 years old in both gender;
8. Weighing of ≥45kg and ≤90kg;
9. Adequate vision and hearing ability to complete all study tests;
10. With a stable caregiver.
11. Informed consent, signed informed consent by legal guardian.

Exclusion Criteria:

1. Have cognitive impairment caused by other types of dementia, mix dementia, Alzheimer's disease(Medial temporal atrophy scale (MTA) score is ≥1.5 (adjusted by age: 65-74 years ≥ 1.5, 75-84 years ≥ 2.0) at baseline MRI screening),frontotemporal dementia, Parkinson's disease dementia, Lewy body dementia, Huntington's disease, etc;
2. Subdural hematoma, traffic hydrocephalus, brain tumor, thyroid disease,vitamin deficiency or other diseases which can lead to cognitive impediment;
3. mood disorders, like depression disorder (HAMD≥17) or anxiety disorder (HAMA≥12);
4. Subject can't complete related test due to severe neurologic deficits, such as hemiplegia, aphasia, audio-visual disorder and so forth;
5. Severe cardiovascular disease(severe arrhythmia, myocardial infarction within 3 months, New York Heart Association Functional Classification III-IV, systolic pressure≥180mmHg or ≤90mmHg);
6. Severe liver or kidney dysfunction, alanine aminotransferase or aspartate transaminase is more than 1.5 times the upper limit of normal, or serum creatinine is more than the upper limit of normal;
7. Uncontrolled diabetes(glycosylated hemoglobin is more than 10%);
8. Asthma, chronic obstructive pulmonary disease, multiple neuritis, myasthenia gravis and muscle atrophy;
9. Severe indigestion, gastrointestinal obstruction, gastric and duodenal ulcers and other gastrointestinal disorders that can affect drug absorption;
10. A medical history of epileptic history, glaucoma, alcoholism, or psycho-substance abuse;
11. History of taking cholinesterase inhibitors, memantine, or proprietary Chinese medicines with clear nootropic effects for the last 1 month;
12. Have taken medications (e.g., antidepressants, benzodiazepines) that affect the central nervous system (CNS), except those for AD, less than 4 weeks；
13. History of hypersensitivity to the treatment drugs;
14. Participate in other clinical study for the last 1 month;
15. Have metal (ferromagnetic) implants, or a cardiac pacemaker and other conditions that make MRI scan not applicable;
16. Or any other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Vascular Dementia Assessment Scale-cognitive subscale(VADAS-Cog) | Baseline, 12-week, 24-week and 36-week.
  Change from baseline to end of double-blind treatment of VADAS-Cog. VADAS-cog is a revision of the ADAS-cog to be a better measure in vascular conditions, and a higher score indicates higher impairment. In addition to ADAS-cog, the VADAS-cog comprises additional frontal lobe tests reflecting attention, working memory, executive function, and verbal fluency.
Clinical Dementia Rating-Sum of Boxes (CDR-SB) | Baseline, 12-week, 24-week and 36-week.
  Change from baseline to end of double-blind treatment of CDR-SB.The CDR-SB is a standard for disease grading in clinical studies of dementia and is used for overall endpoint assessment in clinical trials. It comprehensively assesses the cognitive and functional aspects of dementia patients, including memory, orientation, judgment and problem-solving skills, social affairs, family and hobbies, and personal cooking. The CDR-SB scores from 0 to 18 points, and a higher score indicates higher impairment.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Baseline, 12-week, 24-week and 36-week.
  Change from baseline to end of double-blind treatment of MMSE. MMSE was used to evaluate global cognition, The maximum score for the MMSE is 30, lower score means severe impairment.
Clock drawing test (CDT) | Baseline, 12-week, 24-week and 36-week.
  The changes of the CDT from baseline after 36 weeks treatment. Executive function is assessed by CDT, the maximum score of CDT is 4 points.
Activities of daily living (ADL) | Baseline, 12-week, 24-week and 36-week.
  Change from baseline to end of double-blind treatment of ADL. ADL scale is used to measure the physical self-maintenance ability and instrumental activities of daily living ability.
Delayed story recall (DSR) | Baseline, 12-week, 24-week and 36-week.
  Change from baseline to end of double-blind treatment of DSR. DSR is used to eveluate the memory function, which scores range from 0 to 56.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- dongzhimmen Hospital, Beijing University of Chinese medicine, Beijing, Beijing Municipality, China